CLINICAL TRIAL: NCT01994525
Title: Phase 1 Trial With Challenge to Assess the Safety and Biomarkers of Protection in Malaria-naïve Adults of Immunization Via Mosquito Bite With Radiation-Attenuated Plasmodium Falciparum Sporozoites (IMRAS)
Brief Title: Immunization Via Mosquito Bite With Radiation-attenuated Sporozoites
Acronym: IMRAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Seattle Children's Hospital (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-12-22
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Human Challenge Trials as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1: PfRAS-infected (Experimental): 5 doses (immunizations) of approximately 200 infectious bites (200-400 bites total) from PfRAS-infected mosquitoes (true-immunization). The target dose is 960 infectious bites.
  Challenge occurs 3 weeks after final immunization.
  Interventions: Biological: PfRAS; Other: Challenge
- Cohort 1: Noninfected (Placebo Comparator): Placebo immunization. 5 doses of approximately 200 noninfected bites (200-400 bites total) from irradiated uninfected mosquitoes (mock-immunization). The target dose is 960 noninfected bites.
  Challenge occurs 3 weeks after final immunization.
  Interventions: Biological: Placebo; Other: Challenge
- Cohort 1: Nonimmunized (Other): No protective intervention given.
  Challenge occurs directly after screening.
  Interventions: Other: Challenge
- Cohort 2: PfRAS-infected (Experimental): 3 to 7 doses (immunizations) of approximately 200 infectious bites (200-400 bites total) from PfRAS-infected mosquitoes (true-immunization). The target dose is dependent on protection results in cohort 1.
  Challenge occurs 3 weeks after final immunization.
  Interventions: Biological: PfRAS; Other: Challenge
- Cohort 2: Noninfected (Placebo Comparator): Placebo. 3 to 7 doses of approximately 200 noninfected bites (200-400 bites total) from irradiated, uninfected mosquitoes (true-immunization). The target dose is dependent on protection results in cohort 1.
  Challenge occurs 3 weeks after final immunization.
  Interventions: Biological: Placebo; Other: Challenge
- Cohort 2: Nonimmunized (Other): No protective intervention given.
  Challenge occurs directly after screening.
  Interventions: Other: Challenge
- Hyperimmunity PfRAS-infected (Experimental): Cohort 1 sub-cohort
  3 doses (immunizations) of approximately 200 infectious bites (200-400 bites total) from PfRAS-infected mosquitoes. This arm will receive the first 3 immunizations of Cohort 2.
  Challenge occurs at the same time as Cohort 2 (3-20 weeks after the final immunization)
  Interventions: Biological: PfRAS; Other: Challenge

INTERVENTIONS:
Biological: PfRAS — Radiation-attenuated Plasmodium falciparum sporozoites (PfRAS) administered by the bite of infected Anopheles stephensi mosquitoes
  Other Names: True-immunization; PfRAS infected Anopheles stephensi mosquitoes
  Arms: Cohort 1: PfRAS-infected; Cohort 2: PfRAS-infected; Hyperimmunity PfRAS-infected
Biological: Placebo — Administered by the bite of noninfected Anopheles stephensi mosquitoes
  Other Names: Mock-immunization; Noninfected Anopheles stephensi mosquites
  Arms: Cohort 1: Noninfected; Cohort 2: Noninfected
Other: Challenge — 5 infectious Anopheles stephensi mosquito bites carrying infectious Plasmodium falciparum sporozoites within a controlled clinical environment.

SUMMARY:
This study is to assess the safety, tolerability, and biomarkers of protection in healthy malaria-naïve adults, who will receive bites from Anopheles stephensi mosquitoes either infected with Plasmodium falciparum Sporozoites (PfRAS) (true-immunization) or noninfected (mock-immunization).

DETAILED DESCRIPTION:
This is a Phase 1 open-labeled study. In addition to safety and tolerability of Plasmodium falciparum Sporozoites (PfRAS), this study is a comprehensive, systems biology-based effort to identify and validate biomarkers of protection with PfRAS immunization, comparing sterility protected to nonprotected study subjects. The goal of the trial design is to achieve approximately 50% sterile protection in order to facilitate the identification of biomarkers and correlates of protection.

Following true-immunization or mock-immunization, study subjects and nonimmunized infectivity controls will receive a challenge via the bites of 5 An stephensi mosquitoes carrying infectious P falciparum sporozoites within a controlled clinical environment (controlled human malaria infection, CHMI) to determine the level of sterile protection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant, non-breastfeeding female) 18-50 years of age (inclusive).
* Available and willing to participate for duration of study.
* Able and willing to provide written informed consent.
* Able to complete an Assessment of Understanding with a score of at least 70% correct.
* In good general health with no clinically significant health problems as established by medical history, physical exam and laboratory screening.
* Females of childbearing potential must have a negative pregnancy test at screening and agree to not become pregnant or breastfeed for the duration of the study. She must be willing to use a reliable form of contraception during the study. Reliable forms of birth control include use of condoms, diaphragm or cervical cap, birth control pills, IUD or sperm killing products.
* Agree to refrain from blood donation (except as required in this study) for 3 years following P falciparum challenge.
* Agree not to travel to a malaria-endemic region during the study.
* Good peripheral venous access.

Exclusion Criteria:

* Positive HIV, HBsAg, or HCV serology.
* Positive sickle cell screening test, including evidence of sickle trait.
* Reactivity by CSP or AMA1 ELISpot assay or ELISA as determined by IMRAS Study Specific Procedure #204.
* Anemia (below normal reference laboratory value of hemoglobin) on screening.
* Weight less than 110 pounds (this does not apply to infectivity controls as it is a weight cut-off for subjects undergoing leukapheresis procedure)
* Any history of malaria infection or travel to a malaria endemic region within 6 months prior to first immunization.
* History of long-term residence (> 5 years) in area known to have significant transmission of Pf [cumulative lifetime exposure].
* Use of systemic immunosuppressant pharmacotherapy for greater than 10 days within 60 days of scheduled first immunization (inhaled and topical steroids are allowed; short duration or tapered corticosteroid regimens of 10 days or less that have been discontinued prior to first immunization are allowed).
* Current significant medical condition (cardiovascular, hepatic, renal, pulmonary, or hematological) or evidence of any other serious underlying medical condition identified by medical history, physical examination, or laboratory examination (includes bleeding disorders).
* Plan for surgery between enrollment and day 28 post-challenge (minor procedures, elective corrective vision surgery, and dental procedures are allowed).
* Receipt of immunoglobulin and/or any blood products within 90 days of scheduled leukapheresis or immunization. Version 13.0 (08May2015) 70 US Government Proprietary Deleted: 8 Deleted: 08JULY2014
* Has evidence of increased cardiovascular disease risk (defined as > 5%-10%, 5-year risk) as determined by the method of Gaziano (2008). Risk factors include sex, age (years), systolic blood pressure (mm Hg), smoking status, body mass index (BMI, kg/m2), reported diabetes status, and blood pressure.
* An abnormal electrocardiogram (ECG), defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
* History of a splenectomy.
* History of any other illness or condition that, in the investigator's judgment, may substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives. This may include psychiatric disorders (such as personality disorders, anxiety disorders, or schizophrenia) or behavioral tendencies (including active alcohol or drug abuse) discovered during the screening process that in the opinion of the investigator would make compliance with the protocol difficult.
* History of anaphylactic or severe response to mosquito bites, retinal or visual field changes, or known allergy to the antimalarial chloroquine phosphate, which will be used to treat subjects developing malaria after CHMI.
* Participation in any study involving any investigational vaccine or drug within 30 days prior to the screening visit, or plan to participate in another investigational vaccine/drug research during or within 1 month following participation in this study.
* Use or planned use of any drug with antimalarial activity that would coincide with immunization or challenge.
* History of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine.
* Anticipated use of medications known to cause drug reactions with chloroquine or atovaquone-proguanil (Malarone) such as cimetidine, metoclopramide, antacids, and kaolin during the day 7 to 28 post-challenge period.
* Any other significant findings which, in the investigator's judgment, may substantially increase the risk associated with the subject's participation in the study or compromise the scientific objectives.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events | 7 days
  Occurrence of solicited adverse events (AE) from administration of study immunization (PfRAS)
Unsolicited adverse events | 14 days
  Occurrence of unsolicited adverse events (AEs) from administration of immunization (PfRAS)
Laboratory adverse events | 7 days
  Occurrence of laboratory AEs from administration of study immunization (PfRAS)
Serious adverse events | 52 weeks
  Occurrence of serious adverse events (SAEs) from administration of immunization (PfRAS)
Signs and symptoms related to malaria infection | 7 days
  Occurrence of signs and symptoms related to malaria infection starting 7 days post-Controlled Human Malaria Infection (CHMI) (these will not be recorded as adverse events because they are expected as a result of malaria infection)
Parasitemia | 52 weeks
  Development of parasitemia and time to parasitemia after malaria challenge

SECONDARY OUTCOMES:
Identify and validate immunological PBMC biomarkers | 52 weeks
  Compare Peripheral Blood Mononuclear Cell(s) (PBMC) read-outs between protected and nonprotected subjects and between immunized and mock-immunized subjects.
Identify and validate immunological serum biomarkers | 52 weeks
  Compare serum read-outs between protected and nonprotected subjects and between immunized and mock-immunized subjects.
Identify and validate whole blood immunological biomarkers | 52 weeks
  Compare whole blood read-outs between protected and nonprotected subjects and between immunized and mock-immunized subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Nimfa Teneza-Mora, MD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Naval Medical Research Center Clinical Trials Center (CTC), Bethesda, Maryland, United States

REFERENCES:
- [Derived] Oyong DA, Duffy FJ, Neal ML, Du Y, Carnes J, Schwedhelm KV, Hertoghs N, Jun SH, Miller H, Aitchison JD, De Rosa SC, Newell EW, McElrath MJ, McDermott SM, Stuart KD. Distinct immune responses associated with vaccination status and protection outcomes after malaria challenge. PLoS Pathog. 2023 May 17;19(5):e1011051. doi: 10.1371/journal.ppat.1011051. eCollection 2023 May. PMID 37195999
- [Derived] Du Y, Hertoghs N, Duffy FJ, Carnes J, McDermott SM, Neal ML, Schwedhelm KV, McElrath MJ, De Rosa SC, Aitchison JD, Stuart KD. Systems analysis of immune responses to attenuated P. falciparum malaria sporozoite vaccination reveals excessive inflammatory signatures correlating with impaired immunity. PLoS Pathog. 2022 Feb 2;18(2):e1010282. doi: 10.1371/journal.ppat.1010282. eCollection 2022 Feb. PMID 35108339
- [Derived] Sedegah M, Hollingdale MR, Ganeshan H, Belmonte M, Huang J, Belmonte A, Inoue S, Velasco R, Hickey B, Teneza-Mora N, Lumsden J, Reyes S, Banania JG, Reyes A, Guzman I, Richie TL, Epstein JE, Villasante E. IMRAS-Immunization with radiation-attenuated Plasmodium falciparum sporozoites by mosquito bite: Cellular immunity to sporozoites, CSP, AMA1, TRAP and CelTOS. PLoS One. 2021 Aug 20;16(8):e0256396. doi: 10.1371/journal.pone.0256396. eCollection 2021. PMID 34415964
- [Derived] Hickey B, Teneza-Mora N, Lumsden J, Reyes S, Sedegah M, Garver L, Hollingdale MR, Banania JG, Ganeshan H, Dowler M, Reyes A, Tamminga C, Singer A, Simmons A, Belmonte M, Belmonte A, Huang J, Inoue S, Velasco R, Abot S, Vasquez CS, Guzman I, Wong M, Twomey P, Wojnarski M, Moon J, Alcorta Y, Maiolatesi S, Spring M, Davidson S, Chaudhury S, Villasante E, Richie TL, Epstein JE. IMRAS-A clinical trial of mosquito-bite immunization with live, radiation-attenuated P. falciparum sporozoites: Impact of immunization parameters on protective efficacy and generation of a repository of immunologic reagents. PLoS One. 2020 Jun 17;15(6):e0233840. doi: 10.1371/journal.pone.0233840. eCollection 2020. PMID 32555601